CLINICAL TRIAL: NCT05251831
Title: Evaluation of Activated Platelet Rich Plasma Versus Non-Activated Platelet Rich Plasma in Alopecia Areata
Brief Title: Comparative Study Efficacy and Safety of of Activated Versus Non-Activated PRP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Nouh MD, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ahmed HN AA
Record Dates: First submitted 2022-01-02; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Injections, Intradermal; Platelet Count

STUDY DESIGN:
Intervention Model Description: The 40 patients with alopecia areata will be divided into 2 groups:
  Group A: 20 patients will be treated by activated PRP with Calcium chloride (CaCl2). Those patients will be treated with an intradermal injection.
  Group B: 20 patients will be treated by non-activated PRP through intradermal injection
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Activated plasma rich in platelets (Experimental): Group A: patients were treated by intradermal injections of PRP activated with Calcium chloride 10% solution.
  Interventions: Drug: Intradermal injection
- Non- activated plasma rich in platelets (Placebo Comparator): Group B: patients were treated by intradermal injections of PRP without activation.
  Interventions: Drug: Intradermal injection

INTERVENTIONS:
Drug: Intradermal injection — Platelet-rich plasma (PRP) therapy uses injections of a concentration of a patient's own platelets.
  Other Names: Plasma rich in platelets

SUMMARY:
This was comparative prospective study conducted on 40 subjects, diagnosed with alopecia areata of 40 the scalp, carried in a period from February 2020 and March 2021

DETAILED DESCRIPTION:
Alopecia areata is a common recurrent T cell-mediated autoimmune-induced non-scarring hair loss with not fully understood pathogenesis which affects nearly 2% of the general population during lifetime. The course of the disease is unpredictable and currently, no treatment is available for complete cure or prevention. Platelet-rich plasma is an autologous blood-derived product which widely spread in the last decades for the treatment of different dermatological conditions including different hair disorders.

The aim of this work was to evaluate the efficacy and safety of activated platelet-rich plasma in comparison to non-activated platelet-rich plasma in the treatment of alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed clinically and dermatoscopically as Alopecia areata of the scalp (uni- or 50 multilocularis).
2. Age ranged between 18-50 years in both sex.

Exclusion criteria:

1. Previously treated patients.
2. Pregnant women. 3 Patients with hematological disorders.

4. Local infection at the site. 5. Patients with Hemoglobin <10 g/dL and Platelet count <105/µL. 6. Patients suffer from chronic and psychiatric diseases. 7.Age below 18years or age above 50 years ago.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Hair length in group A | three months
  PRP as treatment option was in indicating its anti-inflammatory properties. 183 PRP effective in AA through anti-inflammatory mechanisms owing to its ability to suppress Monocyte 184 chemotactic protein-1 and owing to the presence of Transforming growth factor (β1 and β2) as was 185 shown by Amable and El-Sharkavy with coauthors

SECONDARY OUTCOMES:
Hair length in Group B | five months
  confirm that PRP is safe effective and well tolerated by 207 patients treatment modality for Alopecia areata. Beside this such method is cost effective as no need 208 any expensive tools for preparation and can be done in outpatients clinics easily.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed abdelaal, Prof, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aithal GP, Watkins PB, Andrade RJ, Larrey D, Molokhia M, Takikawa H, Hunt CM, Wilke RA, Avigan M, Kaplowitz N, Bjornsson E, Daly AK. Case definition and phenotype standardization in drug-induced liver injury. Clin Pharmacol Ther. 2011 Jun;89(6):806-15. doi: 10.1038/clpt.2011.58. Epub 2011 May 4. PMID 21544079
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008
- [Background] Kuty-Pachecka M. Psychological and psychopathological factors in alopecia areata. Psychiatr Pol. 2015;49(5):955-64. doi: 10.12740/PP/39064. English, Polish. PMID 26688846
- [Background] Li F, Ohnishi R, Yamada Y, Kubota J, Domen K, Yamada A, Zhou H. Carbon supported TiN nanoparticles: an efficient bifunctional catalyst for non-aqueous Li-O2 batteries. Chem Commun (Camb). 2013 Feb 11;49(12):1175-7. doi: 10.1039/c2cc37042e. PMID 23289098
- [Background] Strazzulla LC, Wang EHC, Avila L, Lo Sicco K, Brinster N, Christiano AM, Shapiro J. Alopecia areata: Disease characteristics, clinical evaluation, and new perspectives on pathogenesis. J Am Acad Dermatol. 2018 Jan;78(1):1-12. doi: 10.1016/j.jaad.2017.04.1141. PMID 29241771